CLINICAL TRIAL: NCT03113357
Title: The Effect of Myofascial Release Technique on Headache Intensity,Duration,Frequency and Pressure Pain Threshold in Patients With Cervicogenic Headache
Brief Title: The Effect of Myofascial Release in Patients With Cervicogenic Headache
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Amir Massoud Arab, Amir Massoud Arab, University of Social Welfare and Rehabilitation Science, University of Social Welfare and Rehabilitation Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 931672006
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Cervicogenic Headache
Keywords: myofascial release; cervicogenic headache; pain intensity; exercise therapy; pressure pain threshold
MeSH Terms: conditions — Post-Traumatic Headache; Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release technique (Experimental): Subjects lied down in supine with knee flexion. Therapist seated on a stool at the head of the table. Elbows and supinated forearms on the table. Asked the client to lift their head off the table. Position the tips of the first three fingers into the soft tissue immediately inferior to the arc of atlas. The fingers are stabilized in a flexed position - around 45° at the MP and PIP joints. The subject is asked to rest their head back down so the fingertips are in the sub-occipital soft tissues and the finger pads rest firmly against the inferior aspect of the atlas. Once the position is perceived to be comfortable, a series of soft tissue responses will occur, characterized by local softening sensations followed by an increase in the weight of the head.
  Interventions: Other: Myofascial release technique
- conventional exercise therapy (Experimental): Craniocervical flexion exercises, performed in supine lying, aimed to target the deep neck flexor muscles. Then they trained to be able to hold progressively increasing ranges of craniocervical flexion using feedback from an airfilled pressure sensor placed behind the neck. The muscles of the scapula, particularly the serratus anterior and lower trapezius, were trained using inner range holding exercises of scapular adduction and retraction, practiced initially in the prone lying position. The subjects were trained to sit with a natural lumbar lordosis while gently adducting and retracting their scapulas and gently flexed their cranio-cervical spine to facilitate the deep neck flexors.
  Interventions: Other: conventional exercise therapy

INTERVENTIONS:
Other: Myofascial release technique — myofascial release technique take along about 3 minutes. This phase repeated 3 times in each session. At the end, for more release, sub-occipital traction will commence. The subject lies supine with head supported and therapist places the three middle fingers just caudal to the nuchal line, lifts the finger tips upward resting the hands on the treatment table, and then applies a gentle cranial pull, causing a long axis extension. The procedure is performed for 2 to 3 minutes. Subjects in each group received ten physical therapy treatment sessions. Treatment frequency was six times per week for MFR group and every day for exercise group which three times per week have been come to clinical center for checking of exercise by physiotherapist
  Other Names: soft tissue release
  Arms: Myofascial release technique
Other: conventional exercise therapy — All exercises were performed to a count of 7 seconds and subjects were instructed to perform all exercises daily, 15 repetitions each (twice a day). Treatment frequency was every day for exercise group which three times per week have been come to "clinical center" for checking of exercise by physiotherapist. They also could be taught active muscle stretching exercises to address any muscle tightness assessed to be present.
  Arms: conventional exercise therapy

SUMMARY:
Cervicogenic headache (CeH) is a secondary and often unilateral that is known by referring pain from soft or hard cervical structures to occipital, temporal, frontal and sometimes pre-orbital regions. There is higher prevalence of cervical muscle tightness, assessed clinically in CeH patients and anatomically there are some fascial connections between sub-occipital muscles with vertebra of C2 and Dura-mater.Therefore fascial restriction in this region can limit the normal movement of muscles between fascial plates in different directions in sub-occipital region. The purpose of current study was to compare the effect of MFR Technique in the upper cervical region with common (Exs) on pain intensity, frequency, duration and Pressure Pain Threshold (PPT) of upper cervical joints in subjects with CeH.

DETAILED DESCRIPTION:
Cervicogenic headache (CeH) is a secondary and often unilateral that is known by referring pain from soft or hard cervical structures to occipital, temporal, frontal and sometimes pre-orbital regions(Becker, 2010). Its prevalence within the general population is about 0.4-2.5% and in women four times more than men(Racicki, Gerwin, DiClaudio, Reinmann, & Donaldson, 2013). It has been estimated that 15-20% of all chronic headaches include CeH (Racicki et al., 2013). According to reports, at a minimum about 7 million people travail from CeH that cause to waste many daily works and so decrease their performance strongly(Suijlekom, Lamé, Stomp-van den Berg, Kessels, & Weber, 2003). Based on last version of "Cervicogenic Headache International Study Group" a list including some clinical criteria as pain by cervical movement or inappropriate sustained positions, soft tissue stiffness, neck pain and limited cervical Range of Motion (ROM) has been mentioned for CeH. The best available studies has showed that the C2-3 zygapophysial joints are the most common source of CeH, accounting for about 70% of cases(Hall, Briffa, Hopper, & Robinson, 2010; Zito, Jull, & Story, 2006). One of the major problem is overlapping of CeH with other type headaches like migraine and tension type headache (TTH)(Yi, Cook, Hamill-Ruth, & Rowlingson, 2005) but it has been proven that the best clinical test with high sensitivity and specificity for diagnosing of CeH is upper cervical flexion-rotation test (FRT)(Amiri, Jull, & Bullock-Saxton, 2003; Bravo Petersen & Vardaxis, 2015). some investigations have linked CeH to painful dysfunction in the upper three cervical segments (C0-3)(Hall et al., 2007; Ogince, Hall, Robinson, & Blackmore, 2007). Jull and et al at 1999 had noted that there is higher prevalence of cervical muscle tightness, assessed clinically in CeH patients(G Jull, Barrett, Magee, & Ho, 1999; Zito et al., 2006). Nevertheless anatomically, there are some fascial connections between sub-occipital muscles with vertebra of C2 and Dura-mater (Robert Schleip, Jäger, & Klingler, 2012). It has been assumed that fascial limitations in one region of the body cause undue stress in another regions of the body due to fascial continuity, Therefore fascial restriction in this region can limit the normal movement of muscles between fascial plates in different directions in sub-occipital region(Ajimsha, Al-Mudahka, & Al-Madzhar, 2015; Robert Schleip, 2003). Recent Fascia Research Congresses (FRC) explained fascia as a 'soft tissue component of the connective tissue system that percolate the human body(Langevin & Huijing, 2009) and is a part of body tensional force transmission system(R Schleip, Findley, Chaitow, & Huijing, 2012). Myofascial Release (MFR) is a therapeutic technique that uses gentle pressure and stretching (in both forms of direct and indirect approaches) intended to restore decrease pain, optimized length, , and facilitate the release of fascial restrictions caused by injury, stress, repetitive use, and etc (J. F. Barnes, 1990; Robert Schleip, 2003). There are some studies about MFR and its effects that include: increase extensibilities of soft tissues, increase ROM, Improve joint biomechanics, decrease pain and muscles tone significantly (Ajimsha, 2011; Tozzi, Bongiorno, & Vitturini, 2011). Although; a lot of remedies as physiotherapy, electrotherapy, exercises therapy and spinal mobilization are used for cervicogenic headache (GA Jull & Stanton, 2005; Pöllmann, Keidel, & Pfaffenrath, 1997) but it has not been studied specifically about sub-occipital MFR for CeH. Therefor the purpose of current study was to compare the effect of MFR Technique in the upper cervical region with common (Exs) on pain intensity, frequency, duration and Pressure Pain Threshold (PPT) of upper cervical joints in subjects with CeH.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain with referring unilateral pain to sub-occipital region.
* The pain and limitation of C1-C2 rotation with craniocervical FRT.
* Intensifying of Headache by manual pressure to upper cervical muscles and joints.
* Headache frequency of at least one per week a period of previous 6 months

Exclusion Criteria:

* Bilateral headaches (typifying tension headache).
* Intolerance to craniocervical FRT.
* Presence of autonomic system symptoms like vertigo, dizziness and visual impairment.
* Severe specific neck pain as disk herniation, canal stenosis and cervical spondylosis.
* Any condition that might contraindicate myofascial release technique in upper cervical region.
* Physiotherapy for headache in the previous 6 months.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
headache severity | one year
  Pain intensity using Visual Analogue Scale (VAS) were collected at base line and at the end of treatmen

SECONDARY OUTCOMES:
headache frequency | one year
  number of headache days in the past week/month
headache duration | one year
  average number of hours that headaches lasted in the past week
pressure pain threshold | one year
  A pressure threshold algometer was used to measure the pain pressure threshold of a Trigger point of the vastus lateralis muscle before treatment and the end of of transverse and spinous process of C1 and C2 vertebrae before and after 10 treatmen session.

CONTACTS AND LOCATIONS:
Overall Officials: Amir M Arab, professor, Principal Investigator — University of Social Welfare and Rehabilitation Science
Locations (1):
- University of Social Welfare and Rehabilitation Sciences, Tehran, Islamic Republic of, Iran